CLINICAL TRIAL: NCT02242175
Title: Efficacy of Hydrogen Breath Test in the Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2014-0046
Record Dates: First submitted 2014-09-14; First posted 2014-09-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal group (Other)
  Interventions: Device: Glucose breath test (hydrogen breath test)
- irritable bowel syndrome group (Other)
  Interventions: Device: Glucose breath test (hydrogen breath test)

INTERVENTIONS:
Device: Glucose breath test (hydrogen breath test) — Glucose breath test (hydrogen breath test) is the current gold standard for diagnosis of irritable bowel syndrome. Glucose is a sugar that will be broken down by bacteria if present in the small bowel with hydrogen or methane gas as a by-product. The breath sample will be analyzed for hydrogen or methane content to determine if you are able to properly break down the lactose, fructose or sucrose, or if you have bacterial overgrowth.

SUMMARY:
Irritable bowel syndrome is characterized by abdominal discomfort and bowel habit change. It is increasing worldwide. But the pathophysiology of the irritable bowel syndrome is not proven. So, the treatment's target is the relief of the symptoms.

Small intestinal bacterial overgrowth considered as the cause of the irritable bowel syndrome. Because, it is related to the postprandial abdominal discomfort and the abdominal discomfort could be relieved after taking antibiotics. There are several diagnostic methods for small intestinal bacterial overgrowth. hydrogen breath test is non-invasive method for diagnosis of the small intestinal bacterial overgrowth. But, there is no standardized cut-off value for the hydrogen breath test. So, we want to compare the hydrogen breath test between the irritable bowel syndrome patients and normal people. And then, we want to analyze the efficacy of hydrogen breath test for the diagnosis of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. over 19 years old, male and female
2. normal people (control group, who has no abdominal symptoms - diarrhea, constipation etc.)
3. irritable bowel syndrome patients (irritable bowel syndrome means that within the last 3 months abdominal discomfort more than three days for a month and satisfies over the below two items) 1) symptom relived after defecation 2) bowel habit change, the times of defecation changed 3) the change of the morphology of the stool

Exclusion Criteria:

1. patients who do not agree for participation
2. patients who have history for treatment of irritable bowel syndrome
3. patients who is uncontrolled diabetes mellitus
4. patients who have small bowel or large bowel diseases
5. patients who had surgery for abdomen
6. patients who are taking antibiotics, anti-depressants within 1 week
7. patients who are taking proton pump inhibitors or opioids for analgesics
8. patients who have history of bowel adhesion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2014-09; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The difference of H2 elevation level through the hydrogen breath test between the irritable bowel syndrome patients and the normal people | Within the 24 hours after 8-12 hours fasting
  The difference of H2 elevation level through the hydrogen breath test between the irritable bowel syndrome patients and the normal people

SECONDARY OUTCOMES:
The difference of methane level through the hydrogen breath test between the irritable bowel syndrome patients and the normal people | Within the 24 hours after 8-12 hours fasting

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hospital, Seoul, South Korea